CLINICAL TRIAL: NCT06086665
Title: The Real World Efficacy and Safety of Niraparib in Korean Women With Primary and Recurrent Epithelial Ovarian Cancer
Acronym: REFIRM
Status: Completed | Type: Observational
Sponsor: Asan Medical Center (Other)
Collaborators: Samsung Medical Center (Other); Seoul National University Hospital (Other); Severance Hospital (Other); Gangnam Severance Hospital (Other); Keimyung University Dongsan Medical Center (Other); Kyungpook National University Chilgok Hospital (Other); Seoul St. Mary's Hospital (Other); National Cancer Center, Korea (Other Government); Pusan National University Yangsan Hospital (Other); Inje University (Other); Pusan National University Hospital (Other)
Responsible Party: Principal Investigator, Jeong-Yeol Park, MD, PhD, Professor, Asan Medical Center
Other Study IDs: S2022-2461
Record Dates: First submitted 2023-10-11; First posted 2023-10-17 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2026-02

CONDITIONS: Epithelial Ovarian Cancer
MeSH Terms: conditions — Carcinoma, Ovarian Epithelial | interventions — niraparib

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Observation cohort (Cohort A): All patients who did not receive any kind of maintenance therapy for primary epithelial ovarian cancer from Dec 2019 to Dec 2022
- Cohort B: All patients who received or who are receiving niraparib maintenance therapy for primary epithelial ovarian cancer in 1st line setting
  Interventions: Drug: Niraparib
- Cohort C: All patients who received or who are receiving niraparib maintenance therapy for recurrent epithelial ovarian cancer in 2nd or 3rd line setting
  Interventions: Drug: Niraparib
- Cohort D: All patients who received or who are receiving salvage niraparib therapy for recurrent epithelial ovarian cancer in 4th line or more line setting
  Interventions: Drug: Niraparib

INTERVENTIONS:
Drug: Niraparib — Niraparib
  Groups: Cohort B; Cohort C; Cohort D

SUMMARY:
1. To evaluate the efficacy and safety of niraparib in Korean women with primary and recurrent epithelial ovarian cancer who underwent niraparib maintenance therapy
2. To evaluate the efficacy and safety of salvage niraparib therapy in Korean women with heavily pretreated epithelial ovarian cancer.

DETAILED DESCRIPTION:
It has been three years since niraparib was introduced into Korea, and about 600 Korean patients with epithelial ovarian cancer have been treated with this drug. The efficacy and safety of niraparib in primary and recurrent epithelial ovarian cancer were well demonstrated in the NOVA trial and the PRIMA trial, and the efficacy and safety of niraparib in heavily pretreated epithelial ovarian cancer patients were confirmed in the -QUADRA trial. However, safety and efficacy data in Korean women are still scanty. The purpose of this study was to evaluate the safety and efficacy of niraparib in Korean women with primary and recurrent epithelial ovarian cancer.

ELIGIBILITY:
Inclusion Criteria:

* Patients were diagnosed with all histologic type of epithelial ovarian cancer
* Observation cohort (Cohort A): All patients who did not receive any kind of maintenance therapy for primary epithelial ovarian cancer from Dec 2019 to Dec 2022
* Treatment cohort: Epithelial ovarian cancer patients who treated with niraparib as maintenance treatment in any line from Dec 2019 to Dec 2022

  * Cohort B: All patients who received or who are receiving niraparib maintenance therapy for primary epithelial ovarian cancer in 1st line setting
  * Cohort C: All patients who received or who are receiving niraparib maintenance therapy for recurrent epithelial ovarian cancer in 2nd or 3rd line setting
  * Cohort D: All patients who received or who are receiving salvage niraparib therapy for recurrent epithelial ovarian cancer in 4th line or more line setting

Exclusion Criteria:

* Borderline ovarian tumor
* Malignant ovarian germ cell tumor
* Malignant sex-cord stroma tumor
* Other malignancy within 5 years of diagnosis of epithelial ovarian cancer excluding carcinoma in situ of uterine cervix, endometrium, bladder, stomach, papillary thyroid cancer, and non-melanoma skin cancer

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Considering the nature of retrospective study, sample size cannot be calculated based on reference. The investigators have a plan to collect the patient data as much as possible from multi-centers.
Sampling Method: Probability Sample
Enrollment: 850 (Actual)
Dates: Start 2019-12-01 (Actual); Primary Completion 2022-10-31 (Actual); Study Completion 2022-10-31 (Actual)

PRIMARY OUTCOMES:
Progression-free survival | 3 years
  Obtain a survival curve using the Kaplan-Meir method in all cohorts, and compare the survival rates between cohort A vs cohort B in total patients, BRCA WT and mutation patients using the log-rank test. Multivariate survival analysis will be performed using Cox's proportional hazard model.
Safety analysis | 3 years
  The fraction that adverse events occurred, the fraction that dose modification occurred, the fraction that dose delay occurred, and the fraction that treatment discontinuation occurred were calculated, respectively. The comparison of the fractions between groups will be done by the Chi-square test or the Fisher exact test. Comparison of means between groups will be done by Student t test or Mann-Whitney U test.
Overall survival analysis | 3 years
  Obtain a survival curve using the Kaplan-Meir method in all cohorts, and compare the survival rates between cohort A vs cohort B in total patients, BRCA WT and mutation patients using the log-rank test. Multivariate survival analysis is performed using Cox's proportional hazard model.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Obstetrics and Gynecology, University of Ulsan College of Medicine, Asan Medical Center, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-04-11): https://cdn.clinicaltrials.gov/large-docs/65/NCT06086665/Prot_SAP_000.pdf